CLINICAL TRIAL: NCT00168636
Title: The Impact of Different Doses of Vitamin A Supplementation on Male and Female Childhood Morbidity and Mortality
Brief Title: Different Doses of Vitamin A Supplementation and Male and Female Morbidity and Mortality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91096-2dos04; 91096-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Mortality; Morbidity
Keywords: Vitamin A; Mortality; Morbidity; OPV; Sex
MeSH Terms: conditions — Coitus | interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
We previously compared the effect on mortality of the half dose and the full dose currently recommended by WHO. Unexpectedly, the low dose was clearly better for girls, but not for boys. The girls' response might have depended on the last vaccine received before the OPV and VAS campaign. We believe that these findings call for confirmation. In connection with a new campaign, we will examine whether half the dose or the full dose has a more beneficial effect on mortality and morbidity in girls, and furthermore address the potential effect modification by the last vaccine received before the supplementation.

DETAILED DESCRIPTION:
In Guinea-Bissau, a combined OPV and VAS campaign took place in November 2002. Given the uncertainty about the best dose of VAS, we examined whether the half dose compared with the full dose currently recommended by WHO gave an equally good protection against childhood morbidity and mortality. Mortality after supplementation was lower, though not significantly so, for children who had received the half dose. However, there was a highly significant inversion of the effect for boys and girls; while the low dose was clearly better for girls, the full dose might have been slightly better for boys. The girls' responses to the high versus the low dose of vitamin A might have depended on the last vaccine received before the OPV and VAS campaign.

We believe that these findings call for confirmation. In connection with the OPV and VAS campaign in November 2004 in Guinea-Bissau, we intend to examined whether half the dose of the dose currently recommended by WHO as compared to the full dose has a more beneficial effect on mortality and morbidity in girls, and furthermore address the potential effect modification by the last vaccine received before the supplementation.

ELIGIBILITY:
Inclusion Criteria:Between 6 mo and 5 years of age and thus eligible for vitamin A and OPV campaign -

Exclusion Criteria:Overt signs of vitamin A deficiency

-

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11000
Dates: Start 2004-11; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mortality
Morbidity
All outcomes are investigated for interactions between vitamin A, sex, and last vaccine received

SECONDARY OUTCOMES:
Rota infection
Measles infection
Growth

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Yakymenko D, Benn CS, Martins C, Diness BR, Fisker AB, Rodrigues A, Aaby P. The impact of different doses of vitamin A supplementation on male and female mortality. A randomised trial from Guinea-Bissau. BMC Pediatr. 2011 Sep 1;11:77. doi: 10.1186/1471-2431-11-77. PMID 21884606